CLINICAL TRIAL: NCT02501889
Title: Walnut Consumption in a Weight Loss Intervention: Effects on Weight Change, Satiety and Potential Mediating Factors
Brief Title: The Lean Living Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Collaborators: AICR Matching Grant Program (California Walnut Commission and AICR) (Unknown)
Responsible Party: Principal Investigator, Cheryl Rock, Professor, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20154971
Record Dates: First submitted 2015-07-09; First posted 2015-07-17 (Estimated); Last update posted 2017-10-26 (Actual); Status verified 2016-09

CONDITIONS: Overweight and Obesity
Keywords: obesity; overweight; weight loss; satiety; walnuts; gastrointestinal peptides
MeSH Terms: conditions — Overweight; Obesity; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Walnut-rich weight loss diet arm (Experimental): Participants will have an individualized reduced-calorie diet prescription and weight loss counseling session with the project coordinator, who is a registered dietitian. Composition of prescribed diets will be based on individual preferences. During the 6-month intervention, study subjects will participate in individualized counseling and group sessions, with in-person, telephone, email and text message contacts to provide support and behavioral guidance and strategies. All participants will have contact with the project coordinator a minimum of every 1-2 weeks. Walnuts will be provided to participants in the walnut-rich study arm.
  Interventions: Behavioral: Walnut-rich weight loss diet
- Standard weight loss diet arm (Active Comparator): Participants will have an individualized reduced-calorie diet prescription and weight loss counseling session with the project coordinator, who is a registered dietitian. Composition of prescribed diets will be based on individual preferences. During the 6-month intervention, study subjects will participate in individualized counseling and group sessions, with in-person, telephone, email and text message contacts to provide support and behavioral guidance and strategies. Participants assigned to this arm will be instructed to abstain from the consumption of nuts during the study. All participants will have contact with the project coordinator a minimum of every 1-2 weeks.
  Interventions: Behavioral: Standard weight loss diet

INTERVENTIONS:
Behavioral: Walnut-rich weight loss diet — Composition of prescribed diets will be based on individual preferences, with the goal of reduced energy intake and increased energy expenditure. During the 6-month intervention, study subjects will participate in individualized counseling and group sessions, with in-person, telephone, email and text message contacts to provide support and behavioral guidance and strategies. Walnuts will be provided to participants. The overall content of the intervention consists of key elements of cognitive-behavioral therapy for obesity. The physical activity component emphasizes planned aerobic exercise, increased physical activity in the lifestyle, and strength training.
  Arms: Walnut-rich weight loss diet arm
Behavioral: Standard weight loss diet — Composition of prescribed diets will be based on individual preferences, with the goal of reduced energy intake and increased energy expenditure. During the 6-month intervention, study subjects will participate in individualized counseling and group sessions, with in-person, telephone, email and text message contacts to provide support and behavioral guidance and strategies. The overall content of the intervention consists of key elements of cognitive-behavioral therapy for obesity. The physical activity component emphasizes planned aerobic exercise, increased physical activity in the lifestyle, and strength training.
  Arms: Standard weight loss diet arm

SUMMARY:
This study investigates whether walnuts help to promote weight loss, associated with increased meal satiety and satisfaction, in 100 overweight and obese men and women who are participating in a 6-month behavioral weight loss intervention. Participants will be randomly assigned to a walnut-enriched reduced-calorie diet or a standard reduced-calorie diet. Body weight, risk factors for cardiovascular disease, and self-reported feelings relevant to satiety and appetite will be measured at baseline and 3- and 6-month follow-up. Also, the response of gastrointestinal tract hormones following meals with or without walnuts will be measured in a subset of study participants (n=20). Results from this study will contribute to understanding the role of nuts in weight control, including further knowledge of the mechanisms, and will expand knowledge of how nuts in the diet may contribute to the prevention and management of obesity.

DETAILED DESCRIPTION:
Epidemiological studies have linked regular consumption of nuts with lower body mass index and reduced likelihood of weight gain in adulthood. Several mechanisms have been proposed to explain why nuts may facilitate weight management, including their high satiety property which may promote dietary compensation with reduced subsequent energy intake. Although proposed as a possible mediating factor, satiety and satiation in relation to nuts or nut-containing meals have been examined in only a few previous studies. The effects of nut consumption in the context of a weight loss intervention have been examined in only five previously-published randomized studies, which have tested the effects of almonds, pistachios or peanuts (but not walnuts) and have had mixed results.

This project is a study to investigate the effects of a walnut-enriched vs. standard reduced-energy diet on body weight and satiety via pre- and post-meal ratings scales, as well as exploring the response of satiety- and appetite-related gastrointestinal peptides to meals with or without walnuts in a sample subset.

The specific aims of this study are:

1. To compare the effects of a walnut-enriched reduced-energy diet to a standard reduced-energy diet on body weight and cardiovascular disease risk factors in a sample of overweight and obese adults in an intensive 6-month weight loss intervention.
2. To examine whether there is a differential response in satiety- and appetite-related ratings scales in association with a walnut-enriched reduced-energy diet and a standard reduced-energy diet among the participants in this weight-loss study.
3. To examine the response of satiety- and appetite-related gastrointestinal peptides (ghrelin, cholecystokinin, glucagon-like peptide, and peptide YY), to meals with or without walnuts in a sample subset, as an exploratory aim.

The first two aims will be addressed in a randomized controlled study involving 100 overweight or obese men and women assigned to a walnut-enriched reduced-energy diet or a standard reduced-energy diet in the context of a 6-month intensive weight loss intervention. Subjective satiety- and appetite-related ratings will be collected at specific intervals before lunch and dinner using visual analogue scales. Postprandial gastrointestinal peptide response to a meal with or without walnuts, the third and exploratory aim, will be measured in a subset of study participants (n=20) using a within-subject crossover study design.

The investigators hypothesize that participants assigned to the walnut-enriched diet study arm will have greater weight loss and overall better improvements in cardiovascular disease risk factors, and that ratings of hunger, fullness, and anticipated prospective consumption will differ from those of participants assigned to the standard reduced-energy diet. The investigators hypothesize that postprandial satiety- and appetite-related gastrointestinal peptides, which play a role in short-term control of appetite and may be biomarkers of satiety, may differ in response to different isocaloric meal composition. Results from this study will contribute to understanding the role of nuts in weight control, including further knowledge of the explanatory mechanisms, and will expand knowledge of how nuts in the diet may contribute to the prevention and management of obesity.

ELIGIBILITY:
Inclusion Criteria:

* aged 21 years and older
* BMI >27.0 kg/m2 and <40 kg/m2
* non-smoker
* willing and able to participate in clinic visits, group sessions, telephone, and internet communications at specified intervals
* able to provide data through questionnaires and by telephone
* willing to maintain contact with the investigators for 6 months
* willing to allow blood collections
* no known allergy to tree nuts
* capable of performing a simple test for assessing cardiopulmonary fitness

Exclusion Criteria:

* inability to participate in physical activity because of severe disability
* a history or presence of a comorbid diseases for which diet modification and increased physical activity may be contraindicated
* smoker
* self-reported pregnancy or breastfeeding or planning a pregnancy within the next year
* currently actively involved in another diet intervention study or organized weight loss program
* a history or presence of a significant psychiatric disorder or any other condition that, in the investigator's judgement, would interfere with participation in the trial

Ages: 21 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Change in body weight in response to being assigned a walnut-enriched reduced-energy diet or a standard reduced-energy diet in an intensive 6-month weight loss intervention. | 2 years
Change in cardiovascular disease risk factors in response to being assigned a walnut-enriched reduced-energy diet or a standard reduced-energy diet in an intensive 6-month weight loss intervention. | 2 years

SECONDARY OUTCOMES:
Satiety- and appetite-related visual analogue scales in response to being prescribed a walnut- enriched reduced-energy diet or a standard reduced-energy diet among the participants in the weight-loss intervention. | 2 years

OTHER OUTCOMES:
Postprandial blood levels of satiety- and appetite-related gastrointestinal peptides (ghrelin, cholecystokinin, glucagon-like peptide, and peptide YY) following meals with or without walnuts in a sample subset, as an exploratory aim. | 2 years
Satiety- and appetite-related visual analogue scales following meals with or without walnuts in a sample subset, as an exploratory aim. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Cheryl L. Rock, PhD, RD, Principal Investigator — University of California, San Diego
Locations (1):
- UC San Diego, La Jolla, California, United States

REFERENCES:
- [Background] Abazarfard Z, Salehi M, Keshavarzi S. The effect of almonds on anthropometric measurements and lipid profile in overweight and obese females in a weight reduction program: A randomized controlled clinical trial. J Res Med Sci. 2014 May;19(5):457-64. PMID 25097630
- [Background] Alper CM, Mattes RD. Effects of chronic peanut consumption on energy balance and hedonics. Int J Obes Relat Metab Disord. 2002 Aug;26(8):1129-37. doi: 10.1038/sj.ijo.0802050. PMID 12119580
- [Background] Babio N, Toledo E, Estruch R, Ros E, Martinez-Gonzalez MA, Castaner O, Bullo M, Corella D, Aros F, Gomez-Gracia E, Ruiz-Gutierrez V, Fiol M, Lapetra J, Lamuela-Raventos RM, Serra-Majem L, Pinto X, Basora J, Sorli JV, Salas-Salvado J; PREDIMED Study Investigators. Mediterranean diets and metabolic syndrome status in the PREDIMED randomized trial. CMAJ. 2014 Nov 18;186(17):E649-57. doi: 10.1503/cmaj.140764. Epub 2014 Oct 14. PMID 25316904
- [Background] Bes-Rastrollo M, Wedick NM, Martinez-Gonzalez MA, Li TY, Sampson L, Hu FB. Prospective study of nut consumption, long-term weight change, and obesity risk in women. Am J Clin Nutr. 2009 Jun;89(6):1913-9. doi: 10.3945/ajcn.2008.27276. Epub 2009 Apr 29. PMID 19403639
- [Background] Blom WA, Lluch A, Stafleu A, Vinoy S, Holst JJ, Schaafsma G, Hendriks HF. Effect of a high-protein breakfast on the postprandial ghrelin response. Am J Clin Nutr. 2006 Feb;83(2):211-20. doi: 10.1093/ajcn/83.2.211. PMID 16469977
- [Background] Brennan AM, Sweeney LL, Liu X, Mantzoros CS. Walnut consumption increases satiation but has no effect on insulin resistance or the metabolic profile over a 4-day period. Obesity (Silver Spring). 2010 Jun;18(6):1176-82. doi: 10.1038/oby.2009.409. Epub 2009 Nov 12. PMID 19910942
- [Background] Brennan IM, Luscombe-Marsh ND, Seimon RV, Otto B, Horowitz M, Wishart JM, Feinle-Bisset C. Effects of fat, protein, and carbohydrate and protein load on appetite, plasma cholecystokinin, peptide YY, and ghrelin, and energy intake in lean and obese men. Am J Physiol Gastrointest Liver Physiol. 2012 Jul;303(1):G129-40. doi: 10.1152/ajpgi.00478.2011. Epub 2012 May 3. PMID 22556143
- [Background] Casas-Agustench P, Lopez-Uriarte P, Bullo M, Ros E, Gomez-Flores A, Salas-Salvado J. Acute effects of three high-fat meals with different fat saturations on energy expenditure, substrate oxidation and satiety. Clin Nutr. 2009 Feb;28(1):39-45. doi: 10.1016/j.clnu.2008.10.008. Epub 2008 Nov 17. PMID 19010571
- [Background] Delzenne N, Blundell J, Brouns F, Cunningham K, De Graaf K, Erkner A, Lluch A, Mars M, Peters HP, Westerterp-Plantenga M. Gastrointestinal targets of appetite regulation in humans. Obes Rev. 2010 Mar;11(3):234-50. doi: 10.1111/j.1467-789X.2009.00707.x. PMID 20433660
- [Background] Diepvens K, Haberer D, Westerterp-Plantenga M. Different proteins and biopeptides differently affect satiety and anorexigenic/orexigenic hormones in healthy humans. Int J Obes (Lond). 2008 Mar;32(3):510-8. doi: 10.1038/sj.ijo.0803758. Epub 2007 Nov 27. PMID 18345020
- [Background] Foster GD, Shantz KL, Vander Veur SS, Oliver TL, Lent MR, Virus A, Szapary PO, Rader DJ, Zemel BS, Gilden-Tsai A. A randomized trial of the effects of an almond-enriched, hypocaloric diet in the treatment of obesity. Am J Clin Nutr. 2012 Aug;96(2):249-54. doi: 10.3945/ajcn.112.037895. Epub 2012 Jun 27. PMID 22743313
- [Background] Gibbons C, Caudwell P, Finlayson G, Webb DL, Hellstrom PM, Naslund E, Blundell JE. Comparison of postprandial profiles of ghrelin, active GLP-1, and total PYY to meals varying in fat and carbohydrate and their association with hunger and the phases of satiety. J Clin Endocrinol Metab. 2013 May;98(5):E847-55. doi: 10.1210/jc.2012-3835. Epub 2013 Mar 18. PMID 23509106
- [Background] Gibbons C, Finlayson G, Dalton M, Caudwell P, Blundell JE. Metabolic Phenotyping Guidelines: studying eating behaviour in humans. J Endocrinol. 2014 Aug;222(2):G1-12. doi: 10.1530/JOE-14-0020. PMID 25052364
- [Background] Karhunen LJ, Juvonen KR, Flander SM, Liukkonen KH, Lahteenmaki L, Siloaho M, Laaksonen DE, Herzig KH, Uusitupa MI, Poutanen KS. A psyllium fiber-enriched meal strongly attenuates postprandial gastrointestinal peptide release in healthy young adults. J Nutr. 2010 Apr;140(4):737-44. doi: 10.3945/jn.109.115436. Epub 2010 Feb 10. PMID 20147463
- [Background] Kirkmeyer SV, Mattes RD. Effects of food attributes on hunger and food intake. Int J Obes Relat Metab Disord. 2000 Sep;24(9):1167-75. doi: 10.1038/sj.ijo.0801360. PMID 11033986
- [Background] Leidy HJ, Apolzan JW, Mattes RD, Campbell WW. Food form and portion size affect postprandial appetite sensations and hormonal responses in healthy, nonobese, older adults. Obesity (Silver Spring). 2010 Feb;18(2):293-9. doi: 10.1038/oby.2009.217. Epub 2009 Jul 23. PMID 19629055
- [Background] Lejeune MP, Westerterp KR, Adam TC, Luscombe-Marsh ND, Westerterp-Plantenga MS. Ghrelin and glucagon-like peptide 1 concentrations, 24-h satiety, and energy and substrate metabolism during a high-protein diet and measured in a respiration chamber. Am J Clin Nutr. 2006 Jan;83(1):89-94. doi: 10.1093/ajcn/83.1.89. PMID 16400055
- [Background] Li Z, Song R, Nguyen C, Zerlin A, Karp H, Naowamondhol K, Thames G, Gao K, Li L, Tseng CH, Henning SM, Heber D. Pistachio nuts reduce triglycerides and body weight by comparison to refined carbohydrate snack in obese subjects on a 12-week weight loss program. J Am Coll Nutr. 2010 Jun;29(3):198-203. doi: 10.1080/07315724.2010.10719834. PMID 20833992
- [Background] Martinez-Gonzalez MA, Corella D, Salas-Salvado J, Ros E, Covas MI, Fiol M, Warnberg J, Aros F, Ruiz-Gutierrez V, Lamuela-Raventos RM, Lapetra J, Munoz MA, Martinez JA, Saez G, Serra-Majem L, Pinto X, Mitjavila MT, Tur JA, Portillo MP, Estruch R; PREDIMED Study Investigators. Cohort profile: design and methods of the PREDIMED study. Int J Epidemiol. 2012 Apr;41(2):377-85. doi: 10.1093/ije/dyq250. Epub 2010 Dec 20. No abstract available. PMID 21172932
- [Background] Mattes RD, Kris-Etherton PM, Foster GD. Impact of peanuts and tree nuts on body weight and healthy weight loss in adults. J Nutr. 2008 Sep;138(9):1741S-1745S. doi: 10.1093/jn/138.9.1741S. PMID 18716179
- [Background] Mattes RD, Dreher ML. Nuts and healthy body weight maintenance mechanisms. Asia Pac J Clin Nutr. 2010;19(1):137-41. PMID 20199999
- [Background] Mozaffarian D, Hao T, Rimm EB, Willett WC, Hu FB. Changes in diet and lifestyle and long-term weight gain in women and men. N Engl J Med. 2011 Jun 23;364(25):2392-404. doi: 10.1056/NEJMoa1014296. PMID 21696306
- [Background] Natoli S, McCoy P. A review of the evidence: nuts and body weight. Asia Pac J Clin Nutr. 2007;16(4):588-97. PMID 18042516
- [Background] Pelkman CL, Fishell VK, Maddox DH, Pearson TA, Mauger DT, Kris-Etherton PM. Effects of moderate-fat (from monounsaturated fat) and low-fat weight-loss diets on the serum lipid profile in overweight and obese men and women. Am J Clin Nutr. 2004 Feb;79(2):204-12. doi: 10.1093/ajcn/79.2.204. PMID 14749224
- [Background] Rajaram S, Sabate J. Nuts, body weight and insulin resistance. Br J Nutr. 2006 Nov;96 Suppl 2:S79-86. doi: 10.1017/bjn20061867. PMID 17125537
- [Background] Sabate J, Cordero-Macintyre Z, Siapco G, Torabian S, Haddad E. Does regular walnut consumption lead to weight gain? Br J Nutr. 2005 Nov;94(5):859-64. doi: 10.1079/bjn20051567. PMID 16277792
- [Background] Wien MA, Sabate JM, Ikle DN, Cole SE, Kandeel FR. Almonds vs complex carbohydrates in a weight reduction program. Int J Obes Relat Metab Disord. 2003 Nov;27(11):1365-72. doi: 10.1038/sj.ijo.0802411. PMID 14574348
- [Derived] Rock CL, Flatt SW, Barkai HS, Pakiz B, Heath DD. Walnut consumption in a weight reduction intervention: effects on body weight, biological measures, blood pressure and satiety. Nutr J. 2017 Dec 4;16(1):76. doi: 10.1186/s12937-017-0304-z. PMID 29202751